CLINICAL TRIAL: NCT01808742
Title: A Prospective Study Evaluating the Treatment of Forehead and/or Glabellar Lines Utilizing Optimized Algorithms With the Cryo-Touch III Device
Brief Title: Study Evaluating the Treatment of Forehead and/or Glabellar Lines With the CRYO-TOUCH III Device
Status: Completed | Type: Observational
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MYO-0602
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Frown Lines; Glabellar Frown Lines
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Treatment with CryoTouch III device
  Interventions: Device: Treatment with CryoTouch III Device

INTERVENTIONS:
Device: Treatment with CryoTouch III Device — Bilateral forehead treatment with CryoTouch III device on the temporal branch of the facial nerve. Subject will be treated once and may be retreated up to 7 days after initial treatment.

SUMMARY:
myoscience Inc. (Redwood City, CA) has developed a device for a novel, minimally invasive facial rejuvenation procedure designed to soften hyperdynamic facial lines. The myoscience Cryo-Touch III device uses well-established principles of cryobiology to cause localized reduction in muscle activity resulting in a reversible reduction in facial animation and the appearance of facial lines. The device operates on well-established cryobiology principles; that localized exposure to controlled low temperature conditions can alter tissue function. The therapy treats targeted motor nerves with low temperatures via a cold probe in the form of an assembly of small diameter needles, creating a highly localized treatment zone around the probe. The thermal algorithm is designed to produce a reversible loss of nerve conduction resulting in a temporary decrease in muscle contractility. Prior studies of Cryo-Touch, Cryo-Touch II and Cryo-Touch III have provided strong evidence of effectiveness and safety for applications in this indication. The goal of the study described herein is to investigate optimized algorithms and ongoing safety and effectiveness.

DETAILED DESCRIPTION:
The development of facial rhytids or wrinkles is a natural part of the aging process, resulting from the thinning of the dermis and epidermis due to a loss of elastic fibers and collagen and subcutaneous fat loss. Contributors to the formation of facial rhytids include exposure to ultraviolet light (sunlight) and gravity, as well as habitual facial expressions which cause lines to occur in specific facial regions as the skin loses elasticity. In some cases, hyperdynamic activity of underlying facial muscles leads to the development of furrows in the glabella and frontalis areas. Activity of the facial muscles causes hyperdynamic lines independent of the aging process and this can also be undesirable.

With an aging population, the demand for facial rejuvenation techniques has increased. A range of treatment options have been developed to provide reduction in facial lines, including topical medications, neuromuscular inhibiting injections, laser treatments, cosmetic fillers, and surgical facelifts. Those options targeted specifically at hyperdynamic furrows include botulinum toxin injection, injectable fillers, and surgical resection of facial muscles or division of motor nerves. Although botulinum toxin injections have become a popular approach to reduction of glabellar lines by providing partial chemical denervation of the glabellar muscle complex, safety concerns exist related to the use of this toxin. Injectable fillers do not mitigate the underlying muscular activity which produces the facial furrows. Surgical strategies are limited by the risks and complications typically associated with surgery, including bleeding, bruising, scarring, and infection. A non-surgical, minimally invasive approach to elimination of facial hyperdynamic lines which avoids the use of chemical toxins is desirable.

myoscience Inc. (Redwood City, CA) has developed a device for a novel, minimally invasive facial rejuvenation procedure designed to soften hyperdynamic facial lines. The myoscience Cryo-Touch III device uses well-established principles of cryobiology to cause localized reduction in muscle activity resulting in a reversible reduction in facial animation and the appearance of facial lines. The device operates on well-established cryobiology principles; that localized exposure to controlled low temperature conditions can alter tissue function. The therapy treats targeted motor nerves with low temperatures via a cold probe in the form of an assembly of small diameter needles, creating a highly localized treatment zone around the probe. The thermal algorithm is designed to produce a reversible loss of nerve conduction resulting in a temporary decrease in muscle contractility. Prior studies of Cryo-Touch, Cryo-Touch II and Cryo-Touch III have provided strong evidence of effectiveness and safety for applications in this indication. The goal of the study described herein is to investigate optimized algorithms and ongoing safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or Females 30-65 years of age. 2. Forehead wrinkle(s) rating of at least 2 in animation on the 5-point Wrinkle Scale (5WS) which upon physical manipulation of the skin demonstrates a reduction in wrinkle severity.

  3. Glabellar wrinkle score of "1" or higher in animation on the 5-point Glabella Scale (5GS).

  4. Fitzpatrick Skin Type I, II, III or IV. 5. Subject has consented and agreed to participate in all study procedures and visits for the study's duration.

  6. Subject is in good general health, free of any disease state, or physical condition that might impair evaluation of forehead and/or glabellar wrinkle rating or which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* 1. Dermatochalasis with <1mm lid margin when looking straight ahead. 2. Excessive skin laxity. 3. Asymmetry in the upper face. 4. Subjects who actively elevate during a rest cycle. 5. History of facial nerve palsy. 6. Eyebrow or eyelid ptosis. 7. History of neuromuscular disorder. 8. Chronic dry eye symptoms. 9. Allergy or intolerance to lidocaine. 10. Any other clinically significant, in the opinion of the investigator, local skin condition (e.g., skin infection) at target treatment site that may interfere or be a safety concern.

  11. Any physical or psychiatric condition that in the investigator's opinion would prevent adequate study participation.

  12. Chronic medical condition that in the investigator's opinion would affect study participation (such as uncontrolled hypertension, diabetes, hepatitis, HIV, etc.).

  13. Diagnosis of cryoglobulinemia, paroxysmal cold hemoglobinuria, or cold urticaria.

  14. Subject has used aspirin or non-steroidal anti-inflammatory drugs (NSAIDs, e.g., ibuprofen and naproxen) within seven (7) days prior to administration of the device.

  15. Subject has had prior surgery that alters the subcutaneous anatomy of the target treatment sites.

  16. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the investigator.

  17. Subject has undergone another surgical cosmetic procedure or botulinum toxin injection at or above the level of the zygoma (cheekbones) within the past six (6) months prior to administration of the device.

  18. Subject has been treated with fillers (see Section 2.8 Table 1) in the temple or forehead area in the time intervals specified prior to the start of their participation in the study.

  19. Subject has a resting wrinkle score of "2" or higher on the 5WS.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, male or female, age 30 - 65 with forehead and/or glabellar lines deemed significant per protocol inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 30 days
  Wrinkle severity in the target area in animation at 30 days post-treatment as rated by the investigator using the 5-point grading scale.

SECONDARY OUTCOMES:
improvement rating | 56 days
  Changes in from baseline assessments of wrinkle severity based on ratings by the investigator and subject.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Fan, MD, Principal Investigator — 77 Plastic Surgery
Locations (1):
- 77 Plastic Surgery, San Francisco, California, United States